CLINICAL TRIAL: NCT07256834
Title: Incidence of Sore Throat in Postoperative Patients After Use of Betamethasone Gel Compared With Lidocaine Gel During Endotracheal Intubation
Brief Title: Comparison of Efficacy of Betamethasone Gel With Lidocaine Gel in Prevention of Post Endotracheal Intubation Sore Throat.
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jinnah Postgraduate Medical Centre (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: F.2-81/2025-GENL/429/JPMC
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Post Operative Sore Throat at 6hrs and 24hrs After Endotracheal Intubation
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A receiving betamethasone gel during endotracheal intubation (Active Comparator): Group A patients, before induction of anesthesia, endotracheal tube will be lubricated with 2.5ml of 0.05% Betamethasone dipropionate gel, from distal end of cuff to 15cm mark on endotracheal tube
  Interventions: Drug: Betamethasone dipropionate 0.05%
- Group B receiving lidocaine gel during endotracheal intubation (Active Comparator): Group B patients, before induction of anesthesia, endotracheal tube will be lubricated with 2.5ml of 2% Lidocaine gel, from distal end of cuff to 15cm mark on endotracheal tube
  Interventions: Drug: Lidocaine hydrochloride 2%

INTERVENTIONS:
Drug: Betamethasone dipropionate 0.05% — It is corticosteroid indicated for relief of inflammatory and pruritic manifestation
  Arms: Group A receiving betamethasone gel during endotracheal intubation
Drug: Lidocaine hydrochloride 2% — It is amide local anesthetic used for lubrication and pain prevention as topical anesthetic regimen
  Arms: Group B receiving lidocaine gel during endotracheal intubation

SUMMARY:
The goal of this clinical trial is to compare the incidence of postoperative sore throat in adult patients of either gender belonging to ASA I or II ,undergoing endotracheal intubation using betamethasone gel versus lidocaine gel. It aims to determine

1: Difference in efficacy of Betamethasone gel and lidocaine gel in prevention of post operative sore throat after endotracheal intubation.

Patients will be assessed for the presence of a sore throat at 6 hours and 24 hours postoperatively. The severity of the sore throat will be graded using the Post-Operative Sore Throat (POST) score.

DETAILED DESCRIPTION:
This study aims to resolve the debate over the superiority of betamethasone versus lidocaine in preventing POST. Achieving clarity on this issue will not only reduce patient morbidity but also help decrease the duration of hospital stays and lower hospital bed occupancy.The study will commence following the approval of the synopsis by the Research Department of the College of Physicians and Surgeons, Pakistan (CPSP). All patients scheduled for elective surgery under general anesthesia who fulfil the inclusion criteria will be included in the study from Jinnah Postgraduate Medical Center (JPMC). Informed written consent will be obtained from the patients prior to their inclusion in the study.

Initial data, including name, date of presentation, age, weight, height, BMI and gender will be recorded on a predesigned proforma. Patients will then be divided into two group (A and B) through simple random sampling software. In Group A patients, before induction of anesthesia, endotracheal tube will be lubricated with 2.5ml of 0.05% Betamethasone dipropionate gel, from distal end of cuff to 15cm mark on endotracheal tube. In Group B patients, lubrication will be done in a similar manner using 2.5ml of 2% Lidocaine gel. After induction of anesthesia (with IV Propofol 2.5mg/kg, Nalbuphine 0.1mg/kg, Atracurium 0.5mg/kg) and 3 minutes of bag mask ventilation, trachea will be intubated with endotracheal tube of size 7 or 7.5mm according to internal diameter of trachea. Successful endotracheal intubation will be confirmed by capnography and bilaterally equal air entry. Maintenance of general anesthesia will be done by Isoflurane and 60% oxygen mixed with compressed air. Upon completion of surgery, Isoflurane will be discontinued, and residual neuromuscular blockage will be antagonized by Neostigmine 0.05mg/kg. The trachea will be extubated after the patient is fully awake. All patients will be shifted to post-anesthesia care unit where standard ASA monitoring will be continued by a team of anesthetists. The presence and grading of Postoperative sore throat will be done by researcher himself, according to POST Scores at 6 and 24 hours postoperatively, in presence of consultant anesthetist of 5 years of experience. The study will be relevant and specific towards its objective and proper exclusion criteria will be used to control any bias / confounders.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-60 years
2. Either gender
3. ASA I to II
4. Patients planned for elective surgery under general anesthesia not lasting more than 4 hours.

Exclusion Criteria:

1. Patients requiring more than 2 attempts for successful intubation
2. Patients undergoing surgeries of oral cavity or pharynx
3. Mallampati Score of 3 or 4
4. Patients with upper respiratory tract infection
5. Patients already taking steroids
6. Use of nasogastric tube perioperatively

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-22 (Estimated); Primary Completion 2025-12-06 (Estimated); Study Completion 2025-12-06 (Estimated)

PRIMARY OUTCOMES:
Post operative sore throat | Sore throat after endotracheal intubation at 6 hrs and 24hrs post operatively. Sample completion in 2 weeks
  Comparing presence and grading of sore throat in both arms after endotracheal intubation.